CLINICAL TRIAL: NCT07392957
Title: A Phase IB/II Open-label Study of the Safety and Preliminary Efficacy of CTX-009 Administered Either as a Monotherapy or in Combination With CTX-471 in Patients With Recurrent Glioblastoma
Brief Title: Safety and Efficacy of CTX-009 With or Without CTX-471 for Recurrent Glioblastoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-x464
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: VEGF; 4-1BB; CD137; glioblastoma; immunotherapy; targeted therapy; CTX-009; CTX-471
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: After completion of enrollment to Arm 1 (phase IB and phase II), enrollment will open to Arm 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Phase IB Arm 1: CTX-009 monotherapy (Experimental): CTX-009 will be given intravenously at the assigned dose level on an outpatient basis every 2 weeks of a 28-day cycle.
  Interventions: Drug: CTX-009
- Phase IB Arm 2: CTX-009 and CTX-471 combination therapy (Experimental): CTX-009 will be given intravenously at the dose determined to be the recommended phase II dose (RP2D) in Arm 1 every 2 weeks, and CTX-471 will be given intravenously at a dose of 0.3 mg/kg every 2 weeks (day 1 and day 15). On days when both drugs are given, CTX-009 will be given first, followed by a 30-minute observation period, followed by CTX-471. Cycles will be 28 days.
  Interventions: Drug: CTX-009; Drug: CTX-471
- Phase II Expansion Arm 1: CTX-009 monotherapy (Experimental): CTX-009 will be given intravenously at the recommended phase 2 dose (RP2D) determined from Phase IB on an outpatient basis every 2 weeks of a 28-day cycle.
  Interventions: Drug: CTX-009
- Phase II Expansion Arm 2: CTX-009 and CTX-471 combination therapy (Experimental): CTX-009 will be given intravenously at the dose determined to be the recommended phase II dose (RP2D) every 2 weeks (day 1 and day 15). CTX-471 will be given intravenously at a dose of 0.3 mg/kg every 2 weeks (day 1 and day 15). On days when both drugs are given, CTX-009 will be given first, followed by a 30-minute observation period, followed by CTX-471. Cycles will be 28 days.
  Interventions: Drug: CTX-009; Drug: CTX-471

INTERVENTIONS:
Drug: CTX-009 — CTX-009 will be given intravenously over the course of 60 minutes (+/- 5 minutes) on an outpatient basis every 2 weeks of a 28-day cycle.
Drug: CTX-471 — CTX-471 will be given intravenously over the course of 30 minutes (-5/+10) on an outpatient basis every 2 weeks of a 28-day cycle.
  Arms: Phase IB Arm 2: CTX-009 and CTX-471 combination therapy; Phase II Expansion Arm 2: CTX-009 and CTX-471 combination therapy

SUMMARY:
This is a phase IB/II, open-label study evaluating CTX-009 as monotherapy and in combination with CTX-471. The study evaluates the safety and efficacy of the monotherapy and the combination in patients with recurrent glioblastoma. The study tests the hypothesis that treatment with CTX-009 alone or in combination with CTX-471 will lead to enhanced tumor control and prolongation of overall survival of patients with recurrent glioblastoma.

CTX-009 expands on existing anti-angiogenic therapies by ablating key compensatory and resistance mechanisms to bevacizumab, CTX-471 restores local immune reactivity through activation of costimulatory immune mediators. Combination of these two agents may further impair tumor proliferation through synergistic effects on the tumor microenvironment

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiographically confirmed recurrent CNS WHO grade 4 IDH wild-type glioma following standard of care treatment including radiation, chemotherapy, and/or tumor-treating fields. No more than 2 recurrences are allowed.
* At least 18 years of age.
* KPS performance status ≥ 60%
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 75 K/cumm
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN, unless suspected or documented history of Gilbert's Syndrome, in which case ≤ 2.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
  * Urine Protein : Creatinine ratio (UPCR) < 300 mg/g
* The effects of CTX-009 and CTX-471 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 4 months after completion of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Resolution, or stable control with medical management, of all prior anti-cancer therapy toxicities to ≤ grade 1 per NCI-CTCAE v5.0. If the patient has had major surgery, 4 weeks must have elapsed from the date of surgery and the first dose of study drug(s).
* Stable or decreasing dose of corticosteroids and anti-seizure medications for 7 days prior to start of study drug(s). For Arm 2: a maximum of 2 mg daily dose of dexamethasone or equivalent at time of study drug(s) initiation is allowed.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.
* Patients may receive palliative treatment for recurrent disease prior to study enrollment with surgery or laser thermal ablation but must wait at least 4 weeks post-procedure to start study drug(s) and must have recovered from all procedure-related complications.

Exclusion Criteria:

* Have progressed on prior anti-VEGF-A therapy (i.e., bevacizumab) or developed clinically significant adverse reaction to any anti-VEGF therapy (i.e., bevacizumab, regorafenib) which led to discontinuation of treatment. Prior treatment with low dose anti-VEGF therapy for management of symptomatic vasogenic edema or radiation necrosis is permitted as long as progression was not noted while receiving treatment with the anti-VEGF agent, and is not needed for continued control of symptoms. A 4-week washout from last dose of low-dose anti-VEGF therapy is required.
* Prior systemic anti-cancer therapy including: investigational agents or immunotherapy within 4 weeks (can consider 2 week interval for agents with known 5 half-lives <14 days following discussion with study PI); chemotherapy within 4 weeks (6 weeks for BCNU or CCNU); or targeted therapy within 2 weeks prior to treatment.

Note: participants must have recovered from all clinically significant AEs due to previous therapies to ≤ grade 1 or baseline. This does not include AEs deemed not clinically significant by treating physician (i.e., alopecia). Participants with endocrine-related AEs ≤ grade 2 requiring treatment or hormone replacement are eligible if controlled (i.e., clinically asymptomatic) on stable dose of replacement therapy.

* Use of aspirin, NSAIDs, or other antiplatelet agents within 7 days of study drug(s) initiation. Regular use (i.e., daily) of these agents should be avoided while on study treatment.
* Use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes within 7 days of study drug(s) initiation. Prophylactic dosing of DOAC, such as apixaban or edoxaban, or LMWH for patency of venous access devices is allowed (preference is given to DOAC over LMWH).
* History of intraparenchymal or subdural hemorrhage. History of hemorrhage-related or gastroenterological disease including active hemorrhage, hemorrhagic diathesis, coagulopathy, or tumor in great arteries. History of clinically significant gastroenterological disease, such as peptic ulcer, GI bleeding, GI or non-GI fistula, perforation, abdominal abscess, percutaneous drains, clinical symptoms and signs of GI obstruction, need for parenteral hydration or nutrition, or inflammatory bowel disease (IBD).
* History of unprovoked high-risk thromboembolic events.
* A history of the following cardiovascular diseases in the past 5 years (a case-by-case evaluation can be considered in consultation with the study PI):

  * Congestive heart failure that corresponds to Class II or a higher class under NYHA classification or < 50% of LVEF
  * Uncontrolled hypertension (140/90 mmHg despite best care including anti-hypertensive medications). White coat hypertension is not exclusionary.
  * Hypertensive crisis or pre-existing hypertensive encephalopathy
  * Pulmonary hypertension
  * Myocardial infarction
  * Uncontrolled arrhythmia
  * Unstable angina
* Significant vascular diseases (e.g., aortic aneurysm requiring surgery or recent peripheral artery thrombosis) within 6 months prior to study entry
* For Arm 2: Prior treatment with other investigational immune-oncology therapies targeting CD137 (4-1BB).
* For Arm 2: Systemic therapy with non-steroidal immunosuppressive agents within 7 days prior to first dose. Patients with a prior history of autoimmune disease not requiring immunosuppressive therapy may be eligible following discussion with the study PI. Topical, intranasal, intraocular, or inhaled corticosteroids and physiologic replacement for patients with adrenal insufficiency are allowed.
* Prior solid organ or hematologic cell transplantation.
* For Arm 2: Has received a live or live-attenuated vaccine within 30 days prior to the first dose. Note: administration of killed vaccines is allowed.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to CTX-009 or CTX-471.
* Active uncontrolled seizure disorder.
* Active uncontrolled intercurrent illness including, but not limited to: infection, hypertension, open wound(s), or cardiac arrhythmia. Chronic illnesses controlled (i.e., clinically asymptomatic) with oral medications are allowed.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose for Arm 1 or 72 hours of first dose for Arm 2.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase IB Arm 1: Toxicity as measured by number of participants with adverse events | Start of treatment through 60 days after treatment (estimated to be 14 months)
  Adverse events will be graded according to CTCAE v5.0
Phase IB Arm 1: Recommended Phase 2 Dose (RP2D) | Start of treatment through completion of cycle 1 (each cycle is 28 days)
  RP2D will be determined from the phase IB portion of Arm 1 by assessing tolerability. Tolerability is defined as ≤1 among patients experiencing excessive dose limiting toxicities (DLTs). The dose level in phase IB determined to be tolerable is the RP2D.
Phase IB Arm 2: Toxicity as measured by number of participants with adverse events | Start of treatment through 60 days after treatment (estimated to be 14 months)
  Adverse events will be graded according to CTCAE v5.0
Phase II Arm 1: Overall survival rate at 12 months (OS12) | 12 months
  Overall survival is defined from time of treatment start to time of death due to any cause or latest follow-up, whichever is earlier, with an inference focus on 12-month overall survival.
Phase II Arm 2: Overall survival rate at 12 months (OS12) | 12 months
  Overall survival is defined from time of treatment start to time of death due to any cause or latest follow-up, whichever is earlier, with an inference focus on 12-month overall survival.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Start of treatment to end of treatment (estimated total time to be 12 months)
  Overall Response Rate (ORR) is measured as the proportion of patients with complete response (CR) or partial response (PR) as defined by the RANO Response criteria.
  CR is defined as disappearance of all enhancing measurable and non-measurable disease for at least 4 weeks, no new lesions, stable or improved non-enhancing (T2/FLAIR) lesions, off corticosteroids and stable or improved clinically. PR is defined as ≥ 50% decrease of all measurable enhancing lesions for at least 4 weeks, no progression of non-measurable disease, stable or improved non-enhancing (T2/FLAIR) lesions, corticosteroid dose no greater than dose at time of baseline scan, stable or improved clinically
Duration of response (DoR) | Start of treatment to disease progression/recurrence (estimated total time to be 36 months)
  DoR is defined as time from Day 1 of study treatment (CTX-009 with our without CTX-471) to disease progression or death in patients who achieve a complete response (CR) or partial response (PR) as defined by the RANO criteria.
  CR is defined as disappearance of all enhancing measurable and non-measurable disease for at least 4 weeks, no new lesions, stable or improved non-enhancing (T2/FLAIR) lesions, off corticosteroids and stable or improved clinically. PR is defined as ≥ 50% decrease of all measurable enhancing lesions for at least 4 weeks, no progression of non-measurable disease, stable or improved non-enhancing (T2/FLAIR) lesions, corticosteroid dose no greater than dose at time of baseline scan, stable or improved clinically.
  .
Median progression-free survival (mPFS) | Start of treatment to disease progression (estimated to be 36 months)
  mPFS is defined as the time of treatment start to the event of disease progression. Disease progression is measured based on the RANO criteria.
Median overall survival (mOS) | Start of treatment through completion of follow up or death (estimated to be 36 months)
  mOS is measured as the amount of time from treatment start to death due to any cause or latest follow up, whichever is earlier.
Progression free survival at 9 months (PFS9) | 9 months
  PFS9 is measured as amount of time from the start of treatment to the event of disease progression. Disease progression is measured based on the RANO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tanner M Johanns, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared that underlie the results reported (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu